CLINICAL TRIAL: NCT03335592
Title: Cost of Off-label Antibiotics in Osteoarticular Infections: Prospective Study Over 2 Years in a Reference Center for the Management of Complex Bone and Joint Infection
Brief Title: Cost of Off-label Antibiotics in Osteoarticular Infections
Status: Terminated | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Research Assistant, Hospices Civils de Lyon
Other Study IDs: 17-203
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bone Infection; Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the emergence of multidrug-resistant micro-organisms in patients with bone and joint infection (BJI), the prescription of off-labeled antibiotics seem to be more and more common as part of routine care. These new antibiotics are, however, more expensive, and there are no precise data in France regarding the volume and cost of such off-label prescriptions in hospital, in the post-acute care structures, and in the outpatient setting.

The objective of this study is to estimate the cost of using these antibiotics over 2 years for patients in a reference center for the management of complex bone and joint infection (CRIOAc)

ELIGIBILITY:
Inclusion Criteria:

- Patients having had off-label antibiotics between 2014 and 2015 to treat bone and/or joint infection, with or without implant and managed at the CRIOAc Lyon

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having had off-label antibiotics to treat bone and/or joint infection, with or without implant
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Estimation of the cost of the off-label antibiotics | 50 days
  The molecule concerned are: daptomycin, ertapenem, linezolid, ceftaroline, tigecycline and / or colimycin.
  The characteristics of the patients, the type of bone and joint infection and the prescribing methods (dosage, duration) were collected throughout the care path (hospitalization in surgery and / or medicine at CRIOAc or in peripheral hospitals, in post-acute care structure and in the home).
  The duration of dispensation is about 50 days.
  Overall costs for off-label prescriptions were estimated taking account of variations in purchase price invoiced to the reference center.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence des Infections Ostéo-Articulaires complexes (CRIOAc Lyon), Lyon, France

IPD SHARING:
Plan to Share IPD: No